CLINICAL TRIAL: NCT00760422
Title: Clinical Evaluation of NIR (Non-Invasive Infrared) Thermometer Performance
Acronym: NIR
Status: Completed | Type: Observational
Sponsor: Medisim Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 26-115-25
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2008-08

CONDITIONS: Elevated Temperature
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- With fever
  Interventions: Device: NIR
- Without fever
  Interventions: Device: NIR

INTERVENTIONS:
Device: NIR — Thermometer

SUMMARY:
The study is conducted in order to evaluate the performance of the NIT thrmometer by comparing the predictive measurement to equilibrium measurement and to make a final tuning to the thermometer algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Children 0-18 years old, with or without fever that arrive at the unit of emergency medicine in Schneider medical center.
* An informed Consent was signed by the patient or his guardian.

Exclusion Criteria:

* The medical stuff decides that the patient can't participate.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 500 patients from both genders, 0-18 years old
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel